CLINICAL TRIAL: NCT04619420
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study With a Long-Term Extension Treatment Period to Assess the Efficacy and Safety of JNJ-63733657, an Anti-tau Monoclonal Antibody, in Participants With Early Alzheimer's Disease
Brief Title: A Study of JNJ-63733657 in Participants With Early Alzheimer's Disease
Acronym: Autonomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108832; 63733657ALZ2002 (Other: Janssen Research & Development, LLC); 2020-000116-30 (EudraCT Number); 2022-501188-42-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Cognitive Dysfunction; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: There will be 3 treatment arms for the Double-Blind treatment period, whereas there will be only 2 treatment arms for the Long-Term extension treatment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- JNJ-63733657 Low-dose (Experimental): Participants will receive single dose of JNJ-63733657 low-dose administered by intravenous (IV) infusion every 4 weeks during the double-blind treatment period. Participants will have an option to continue with the long-term extension (LTE) phase of the trial and will continue to receive the same treatment and dose during the LTE treatment period.
  Interventions: Drug: JNJ-63733657
- JNJ-63733657 High-dose (Experimental): Participants will receive single dose of JNJ-63733657 high-dose administered by IV infusion every 4 weeks during double-blind treatment period. Participants will have an option to continue with the LTE phase of the trial and will continue to receive the same treatment and dose during the LTE treatment period.
  Interventions: Drug: JNJ-63733657
- Placebo (Placebo Comparator): Participants will receive single dose of matching placebo to JNJ-63733657 administered by IV infusion every 4 weeks during double-blind treatment period. Participants will have an option to continue with the LTE phase of the trial and will be re-randomized in a 1:1 ratio to receive either JNJ-63733657 low-dose or JNJ-63733657 high-dose during the LTE treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-63733657 — JNJ-63733657 low or high dose will be administered by IV infusion.
  Arms: JNJ-63733657 High-dose; JNJ-63733657 Low-dose
Drug: Placebo — Placebo matching to JNJ-63733657 will be administered by IV infusion.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effect of JNJ-63733657 versus placebo on clinical decline as measured by the Integrated Alzheimer's Disease Rating Scale (iADRS), a composite of cognition and function.

ELIGIBILITY:
Inclusion Criteria:

* Early Alzheimer's disease (AD): Gradual and progressive subjective decline in the participant's cognition over at least the past 6 months, as reported by the participant and informant (study partner) and Clinical Dementia Rating-Global Score (CDR-GS) of 0.5 and memory box score greater than or equal to (>=) 0.5 at screening
* Participants must have positive tau PET results
* Able to read and write and with a minimum 5 years of formal education as reported by participant and study partner at screening
* Have a designated study partner who has adequate literacy to participate and be judged to have high likelihood of completing the study with the participant
* Male participants must agree not to donate sperm for the purpose of reproduction during the study and up to 16 weeks after receiving the last dose of study intervention

Exclusion Criteria:

* Participants with CDR GS >=2 at predose baseline Clinical Dementia Rating (CDR) administration
* Participants who fulfill diagnostic criteria for Mild Cognitive Impairment (MCI) or dementia/mild or major neurocognitive disorder suspected to be due to any etiology other than AD (example, Parkinson's disease, cerebrovascular disease, normal pressure hydrocephalus, head injury, drug or alcohol abuse/dependence, anoxic brain injury, (Et cetera[etc])
* Geriatric Depression Scale (GDS) 30 score greater than (>) 12
* Hachinski Ischemic Scale (HIS) >4
* Has received medications that affect the central nervous system (CNS), except treatments for AD, for less than 2 months; that is, doses of chronic medications that effect the CNS should be stable for at least 2 months before the start of screening. If a participant has recently stopped a chronic medication that effects the CNS, he or she must have discontinued treatment at least 2 months before the start of screening. Chronic use of benzodiazepines is not permitted

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) Total Score at Week 104 | Week 104
  The linear combination of the ADAS Cog13 and ADCS ADL MCI that serves as a composite of cognition and function (overall clinical status) of the participant and score range from 0 to 138 with lower scores indicating worse performance. The iADRS will be a combination of ADAS Cog13 (score 0 to 85, higher scores indicate worse cognitive performance) and ADCS-ADL MCI (yielding a score 0 to 53, lower scores indicate worse daily function).

SECONDARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale Cognitive subscale 13-item version (ADAS-Cog 13) Total Score at Week 104 | Week 104
  ADAS-Cog11 consists of 11 tasks measuring the disturbances of memory, language, praxis, attention, and other cognitive abilities. The modified ADAS-Cog 13 item scale includes all original ADAS-Cog items with the addition of a number cancellation task and a delayed free recall task, for a maximum total score of 85 points, with higher scores indicative of worse cognitive performance. Thus, a negative change from baseline represents improvement in cognition. Items are recorded on an electronic device which will provide the ADAS-Cog 13 total score.
Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living for Mild Cognitive Impairment (ADCS-ADL MCI) Total Score at Week 104 | Week 104
  ADCS-ADL MCI is a functional measure based on information provided by the study partner (informant) that describes the performance of participants in several ADLs. It assesses 18 instrumental activities of daily living (higher level daily functions) and one basic daily function (dressing). Total score ranges from 0 to 53 with higher scores indicating less impairment.
Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Index Score at Week 88 | Baseline, Week 88
  The RBANS includes 12 subtests that are divided into 5 RBANS indices: 1-Immediate memory (List learning and story memory); 2-Visuospatial/constructional (figure copy and line orientation); 3-Language (picture naming and semantic fluency); 4-Attention (digit span and coding); 5-Delayed memory (list recall, list recognition, story memory, and figure recall) will be reported. Index scores are expressed as an age-adjusted standard score with a normal mean of 100 and an SD of 15. The sum of Index Scores is the sum of the 5 index scores, and the Sum of Index Scores is converted to an RBANS Total Scale Index Score via a mapping table. RBANS Total Scale Index Score is a norm-based t-score, based on a distribution with a mean of 100 and standard deviation (SD) of 15. Higher scores on each sub measure and index indicate better performance.
Change From Baseline in RBANS Indices at Week 88 | Baseline, Week 88
  Change from baseline in RBANS indices will be assessed. The RBANS includes 12 subtests that are divided into 5 RBANS indices: 1-Immediate memory (List learning and story memory); 2-Visuospatial/constructional (figure copy and line orientation); 3-Language (picture naming and semantic fluency); 4-Attention (digit span and coding); 5-Delayed memory (list recall, list recognition, story memory, and figure recall) will be reported.
Change From Baseline in Clinical Dementia Rating- Sum of Boxes (CDR-SB) at Week 104 | Baseline, Week 104
  CDR is a global clinical staging instrument that includes 3 cognitive and 3 functional ratings, including: memory, orientation, judgment and problem solving, involvement in community affairs, home and hobbies, and personal care based on the CDR interview. The CDR is scored 2 ways yielding a global CDR score (CDR GS, derived from an algorithm including categorical scoring of 0, 0.5, 1, 2, and 3), as well as CDR-Sum of Boxes (CDR-SB, the continuous sum of 6 domains, up to a total score of 18, with higher scores representing worse disease state). The Sum of boxes and global score is calculated from the overall CDR.
Change from Baseline in Neuropsychiatric Inventory (NPI) at Week 104 | Baseline, Week 104
  The NPI is a measure of psychobehavioral disturbances, assessing the frequency and severity of disturbances in 12 domains. Frequency for each domain is rated on a 4 point scale (from 1=rarely to 4=very often) and severity on a 3 point scale (from 1=mild to 3=severe), with the score for each domain being the product of the frequency and severity scores, such that each domain is scored from 1 to 12. The NPI total score is the sum of the 12 domain scores, ranging from 0 (best) to 144 (worst).
Percentage of Participants Progressing From Clinical Dementia Rating- Global Score (CDR-GS) 0 to 0.5 or Higher, 0.5 to 1 or Higher, 1 to 2 or Higher, from Baseline to Post-baseline through Week 104 | From Baseline through Week 104
  The CDR is a subjectively rated outcome measure that serves as a global clinical staging instrument that includes 3 cognitive and 3 functional ratings, including: 1) memory, 2) orientation, 3) judgment and problem solving, 4) involvement in community affairs, 5) home and hobbies, and 6) personal care based on the CDR interview. The CDR is scored 2 ways yielding a global CDR score (CDR GS, derived from an algorithm developed by the Knight Alzheimer Disease Research Center at Washington University School of Medicine in St. Louis, Missouri, US, and including categorical scoring of 0= cognitively unimpaired, 0.5= mild cognitive impairment, 1= mild dementia, 2= moderate dementia, and 3= severe dementia), as well as CDR-Sum of Boxes (CDR-SB, the continuous sum of 6 domains, up to a total score of 18, with higher scores representing worse disease state).
Change From Baseline in Brain tau Burden as Measured by tau PET at Week 104 | Baseline, Week 104
  Change from baseline in brain tau burden, as measured by tau positron emission tomography (PET) will be assessed.
Change From Baseline in Cerebrospinal Fluid (CSF) concentrations of Total, Free, and Bound p217+tau Fragments at Week 104 | Baseline, Week 104
  Change from baseline in CSF concentrations of total, free, and bound p217+tau (phosphorylated tau) fragments will be assessed.
CSF Concentrations of JNJ-63733657 | At Weeks 52, 104, 208 (End of Treatment)
  CSF concentrations of JNJ-63733657 will be assessed.
Serum Concentrations of JNJ-63733657 | At Weeks 4, 8, 12, 16, 20, 24, 36, 52, 76, 104, 128, 156, 180, 208, 232 (End of treatment)
  Serum concentrations of JNJ-63733657 will be assessed.
Anti-Drug Antibody to JNJ-63733657 | Up to 245 Weeks (90 days [+-7 days] after last dose of study intervention)
  Anti-drug antibody to JNJ-63733657 will be assessed.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 245 Weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Number of Participants with Treatment-Emergent Adverse Event of Special Interest (AESI) | Up to 245 Weeks
  Number of participants with a treatment-emergent AESI will be reported.
Number of Participants with Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability | Up to 245 Weeks
  An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to 245 Weeks
  Number of participants with ECG abnormalities will be reported.
Number of Participants with Clinical Laboratory Abnormalities | Up to 245 Weeks
  Number of participants with clinical laboratory (hematology, clinical chemistry, and urinalysis) abnormalities will be assessed.
Number of Participants with Physical and Neurological Examination Abnormalities | Up to 245 Weeks
  Number of participants with physical (body weight, height) and neurological (evaluation of mental status, cranial nerves, motor ability [including strength, tone, and involuntary movements], coordination [including finger-to-nose, gait, and postural reflexes], and sensation [including proprioception, cold, light touch, and deep tendon reflexes]) examination abnormalities will be reported.
Percentage of Participants with Vital Sign Abnormalities | Up to 245 Weeks
  Percentage of participants with vital sign abnormalities (temperature, pulse rate, systolic blood pressure [BP], diastolic BP) will be reported.
Changes From Baseline in Brain Magnetic Resonance Imaging (MRI) Safety Findings | Baseline and Up to 4.5 years (End of treatment)
  Changes from baseline in brain MRI safety findings (brain tumors, aneurysm or atrioventricular malformations, territorial stroke (excluding smaller watershed strokes), recent hemorrhage (parenchymal or subdural), or obstructive hydrocephalus) will be assessed.
Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) score | Baseline and Up to 245 Weeks
  C-SSRS is semi structured clinician-administered questionnaire designed to solicit the occurrence, severity, and frequency of suicide-related ideation and behaviors . Total score ranges from 1 to 10, a score of 0 will be assigned (0="no event that can be assessed on the basis of C-SSRS"). Higher scores indicate greater severity. The maximum score assigned for each participant will also be summarized into one of three broad categories: no suicidal ideation or behavior (0), suicidal ideation (1 to 5), suicidal behavior (6 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (122):
- United States (55):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Dignity Health, Phoenix, Arizona
  - Irvine Clinical Research, Irvine, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Pacific Research Network Prn, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research LLC, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of SWFL, Fort Myers, Florida
  - Clinical NeuroScience Solutions Inc, Jacksonville, Florida
  - Alphab Global Research, Jupiter, Florida
  - K2 Medical Research, Maitland, Florida
  - Tandem Intermediate LLC, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Miami Jewish Health System, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Charter Research, The Villages, Florida
  - ClinCloud Clinical Research, Viera, Florida
  - Alzheimers Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology and Premier Research Institute, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Sandhill Research, Decatur, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alexian Brothers Medical Center - Neuroscience Research Institute, Elk Grove Village, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Anil Nair dba Alzheimer's Disease Center, Braintree, Massachusetts
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Velocity Clinical Research, East Syracuse, New York
  - New York University Medical Center, New York, New York
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Lou Revo Center for Brain Health, Cleveland, Ohio
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Keystone Clinical Studies LLC, Plymouth Meeting, Pennsylvania
  - Brown University School of Medicine, Providence, Rhode Island
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Memory Clinic Inc, Bennington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Neuro Trials Victoria, Carlton
  - Austin Health, Ivanhoe
  - HammondCare Neurodegenerative Clinical Trials - VIC, Malvern
  - Australian Alzheimer's Research Foundation Incorporated, Nedlands
  - Royal Melbourne Hospital, Parkville
- Belgium (8):
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - UCL Hopital Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
- Canada (5):
  - Parkwood Institute, London, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - UHN-Toronto Western Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- France (9):
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - Hopital Roger Salengro - CHU Lille, Lille
  - CHU Nantes - Hopital Nord Laënnec, Nantes
  - Hopital Lariboisiere-Fernand Widal, Paris
  - Hopital Pitie Salpetriere, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Hopital Charles Nicolle, Rouen
  - CHU Toulouse - Hôpital La Grave, Toulouse
  - Hôpital Bretonneau, Tours
- Japan (22):
  - Takeda General Hospital, Aizu-Wakamatsu
  - Inage Neurology and Memory Clinic, Chiba
  - Kawashima Neurology Clinic, Fujisawa-shi
  - Fukuoka University Hospital, Fukuoka
  - Keikokai P-One Clinic, Hachiōji
  - Himeji Central Hospital Clinic, Himeji
  - Shonan Kamakura General Hospital, Kamakura-shi
  - National Hospital Organization Hizen Psychiatric Center, Kanzaki-gun
  - Koukan Clinic, Kawasaki
  - Kobe City Medical Center General Hospital, Kobe
  - Rijikai Medical Corporation Katayama Medical Clinic, Kurashiki-shi
  - Kurume University Hospital, Kurume
  - Rakuwakai Otowa Hospital, Kyoto
  - Rakuwakai Otowa Rehabilitation Hospital, Kyoto
  - Saiseikai Narashino Hospital, Narashino
  - National Center For Geriatrics And Gerontology, Obu-shi
  - Clinical Research Hospital Tokyo, Shinjuku-ku
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - Nagomi Clinic, Toyonaka-shi
  - Jinsenkai MI Clinic, Toyonaka-shi
  - Yokohama Brain and Spine Center, Yokohama
- Netherlands (4):
  - BRC - Den Bosch, 's-Hertogenbosch
  - BRC - Amsterdam, Amsterdam
  - QPS Netherlands, Leeuwarden
  - BRC Zwolle, Zwolle
- Spain (9):
  - Centro At. Esp. Oroitu, Algorta - Getxo
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Fund. Ace-Inst. Cat. Neuroc. Aplicades, Barcelona
  - Idc Salud Hosp. Gral. de Catalunya, Barcelona
  - Hosp. Univ. Santa Maria, Lleida
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Univ. I Politecni La Fe, Valencia
- Karolinska Universitetssjukhuset, Stockholm, Sweden
- United Kingdom (2):
  - Royal United Hospital, Bath
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Perez-Ruixo C, Li L, Galpern WR, Perez-Ruixo JJ. Mechanistic Population Pharmacokinetic-Pharmacodynamic Model of the Tau-Targeted Antibody Posdinemab in Healthy Participants and Participants with Alzheimer's Disease. Clin Pharmacol Ther. 2025 Dec 22. doi: 10.1002/cpt.70173. Online ahead of print. PMID 41431125